CLINICAL TRIAL: NCT04397562
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Adaptively Designed Clinical Trial of the Efficacy and Safety of Levilimab (BCD-089) in Patients With Severe COVID-19
Brief Title: A Clinical Trial of the Efficacy and Safety of Levilimab (BCD-089) in Patients With Severe COVID-19
Acronym: CORONA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-089-4
Record Dates: First submitted 2020-05-19; First posted 2020-05-21 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2020-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — levilimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LVL group (Experimental): Single subcutaneous administration of levilimab at a dose of 324 mg in combination with standard therapy
  Interventions: Drug: Levilimab
- Placebo group (Placebo Comparator): Single subcutaneous administration of placebo in combination with standard therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levilimab — Levilimab 324 mg
  Arms: LVL group
Drug: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
The objective: to study the efficacy and safety of levilimab in subjects with severe COVID-19.

DETAILED DESCRIPTION:
This study is multicenter, comparative, randomized, double-blind, placebo controlled clinical trial with adaptive design. Females and males, aged 18 years and older, admitted to hospital with severe COVID-19 pneumonia on SOC therapy will receive either levilimab 324 mg s/c or placebo s/c. In case of no clinical improvement is observed, investigator can administer a rescue therapy - open label LVL 324 mg s/c. The outcomes will be assessed up to day 60. Results of interim analysis of safety and efficacy data of first 60 enrolled subjects will be submitted for independent DMC review and decision about changes to the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent (subject; legally authorized representative) or signed conclusion of panel of independent medical doctors
2. Males and non-pregnant females aged 18 years or older at the IC date
3. Positive test for SARS-CoV2 nucleic acid (RNA) at the IC date
4. Admitted as inpatient to a hospital with radiologically confirmed pneumonia
5. Severe form of COVID-19.
6. Subjects meeting any of the following criteria:

   * Total respiratory rate > 30 breaths per minute
   * SpO2 ≤ 93%
   * PaO2 /FiO2 ≤ 300 mmHg
   * Chest imaging (X-ray, CT, US) showed lesion progression within 24-48 hours >50%
   * Decrease of consciousness level, Psychomotor agitation/irritability
   * Hemodynamically unstable (systolic blood pressure <90 mmHg or diastolic blood pressure < 60 mmHg or urine output < 20 ml/h)
   * Arterial lactate > 2 mmol/l
   * qSOFA (quick sequential organ failure assessment score) > 2. Subjects meeting three following criteria: Low blood pressure (SBP ≤ 100 mmHg); High respiratory rate (≥ 22 breaths/min); Altered mentation (Glasgow Coma Scale ≤ 14)

Exclusion Criteria:

1. Critical COVID-19. Subjects meeting any of the following:

   * Respiratory failure and requiring invasive mechanical ventilation (tracheal intubation)
   * Septic shock
   * Multiple organ failure
2. Life expectancy < 24h, in the opinion of the investigator,
3. Unlikely to remain at the investigational site beyond 48 hours
4. Use of other monoclonal antibodies for COVID-19 treatment
5. Current treatment with immunosuppressive agents (including corticosteroids)
6. Participating in other drug clinical trials at the IC date or within 60 days after randomization (participation in COVID-19 anti-viral trials may be permitted if approved by Sponsor)
7. Laboratory values:

   * ALT / AST > 10 ULN at screening
   * Platelets < 50х109/l at screening
   * Absolute Neutrophil Count < 1х109/l at screening
8. Suspected active bacterial, fungal, viral, or other infection (besides COVID-19)
9. Confirmed active tuberculosis
10. History of allergic reaction to monoclonal antibodies
11. Pregnancy or breastfeeding
12. Any illness or laboratory findings that, in the opinion of the study investigator, might pose an additional risk to the patient by their participation in the study,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with sustained clinical recovery | Day 14
  Sustained clinical recovery is defined as either an improvement of at least 2 categories relative to baseline on a 7-Category Ordinal Scale of Clinical Status or reaching categories "Discharged" / "Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care" at day 14.

SECONDARY OUTCOMES:
Proportion of patients reporting each category of 7-Category Ordinal Scale of Clinical Status | Day 30
  7-Category Ordinal Scale of Clinical Status:
  1. Not hospitalized / Discharged
  2. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  3. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise)
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, requiring non-invasive ventilation or high flow oxygen devices
  6. Hospitalized, requiring invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  7. Death
Proportion of patients transferred to the ICU | Day 60
Duration of fever | Day 60
Duration of hospitalization | Day 60
Change in ESR | Day 30
Change in serum CRP level | Day 30
Change in serum IL-6 level | Day 30

CONTACTS AND LOCATIONS:
Locations (16):
- Russia (16):
  - State Budgetary Healthcare Institution Kaluga region "Kaluga Regional Clinical Hospital", Kaluga
  - State Budget Institution of the Republic of Dagestan "Republican Clinical Hospital", Makhachkala
  - A.N. Bakulev National Medical Research Center of Cardiovascular Surgery, Moscow
  - City Clinical Hospital No. 40 of the Department of Health of the city of Moscow, Moscow
  - City Clinical Hospital No.52, Moscow
  - City Clinical Hospital № 15 named. O.M. Filatov, Moscow
  - City Clinical Hospital №1 named after N.I. Pirogov, Moscow City Health Department, Moscow
  - Federal State Budgetary Institution "Central Clinical Hospital with Clinic", Office of the President of the Russian Federation, Moscow
  - I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow
  - Pirogov Russian National Research Medical University, Moscow
  - Railway clinical hospital named after N.A. Semashko, Moscow
  - Almazov National Medical Research Centre, Saint Petersburg
  - Clinical Infectious Disease Hospital named after S.P. Botkin, Saint Petersburg
  - North-western State Medical University named after I.I.Mechnikov, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "Bashkir State Medical University" of the Ministry of Healthcare of the Russian Federation, Ufa
  - Federal State Budgetary Educational Institution of Higher Education "North Ossetian State Medical Academy" of the Ministry of Health of the Russian Federation (FSBEI HE SOGMA of the Ministry of Health of Russia), Vladikavkaz

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lomakin NV, Bakirov BA, Protsenko DN, Mazurov VI, Musaev GH, Moiseeva OM, Pasechnik ES, Popov VV, Smolyarchuk EA, Gordeev IG, Gilyarov MY, Fomina DS, Seleznev AI, Linkova YN, Dokukina EA, Eremeeva AV, Pukhtinskaia PS, Morozova MA, Zinkina-Orikhan AV, Lutckii AA. The efficacy and safety of levilimab in severely ill COVID-19 patients not requiring mechanical ventilation: results of a multicenter randomized double-blind placebo-controlled phase III CORONA clinical study. Inflamm Res. 2021 Dec;70(10-12):1233-1246. doi: 10.1007/s00011-021-01507-5. Epub 2021 Sep 29. PMID 34586459
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34586459/